CLINICAL TRIAL: NCT02574637
Title: A Phase 2b Double-Blind, Multi-Dose, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MEDI2070 in Subjects With Moderate to Severe Crohn's Disease Who Have Failed or Are Intolerant to Anti-tumor Necrosis Factor-alpha Therapy
Brief Title: Evaluation of Efficacy and Safety of Brazikumab (MEDI2070) in Participants With Active, Moderate to Severe Crohn's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated for business reasons; not due to safety or efficacy concerns.
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D5170C00002; 2015-000609-38 (EudraCT Number)
Record Dates: First submitted 2015-09-24; First posted 2015-10-14 (Estimated); Results first posted 2020-05-15 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Crohn's Disease
Keywords: MEDI2070; inflammatory bowel disease; moderate to severe Crohn's Disease; IL-23
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — MEDI2070

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Placebo-matching brazikumab intravenous (IV) infusion and subcutaneous (SC) injection at Weeks 0 and 4 followed by placebo-matching brazikumab SC injection at Weeks 8 and 12 in the induction phase and at Weeks 16, 20 and 24 in the maintenance phase. Participants received brazikumab 210 mg, SC injection every 4 weeks up to Week 48 in the open-label period.
  Interventions: Drug: Brazikumab IV Infusion; Drug: Brazikumab SC Injection; Drug: Placebo
- Brazikumab High Dose (Experimental): Brazikumab 700 mg, IV infusion and placebo-matching brazikumab, SC injection at Weeks 0 and 4 followed by brazikumab 210 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 210 mg, SC injection every 4 weeks in the maintenance phase and open-label period up to Week 48.
  Interventions: Drug: Brazikumab IV Infusion; Drug: Brazikumab SC Injection; Drug: Placebo
- Brazikumab High-Medium Dose (Experimental): Brazikumab 280 mg, IV infusion and placebo-matching brazikumab, SC injection at Week 0 followed by brazikumab 210 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 210 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 210 mg, SC injection every 4 weeks in the maintenance phase and open-label period up to Week 48.
  Interventions: Drug: Brazikumab IV Infusion; Drug: Brazikumab SC Injection; Drug: Placebo
- Brazikumab Low-Medium Dose (Experimental): Brazikumab 210 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 0 followed by brazikumab 105 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 105 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 105 mg, SC injection every 4 weeks up to Week 24 in the maintenance phase. Participants received brazikumab 210 mg, SC injection, every 4 weeks up to Week 48 in the open-label period.
  Interventions: Drug: Brazikumab IV Infusion; Drug: Brazikumab SC Injection; Drug: Placebo
- Brazikumab Low Dose (Experimental): Brazikumab 70 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 0 followed by brazikumab 35 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 35 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 35 mg, SC injection every 4 weeks up to Week 24 in the maintenance phase. Participants received brazikumab 210 mg, SC injection, every 4 weeks up to Week 48 in the open-label period.
  Interventions: Drug: Brazikumab IV Infusion; Drug: Brazikumab SC Injection; Drug: Placebo

INTERVENTIONS:
Drug: Brazikumab IV Infusion — Brazikumab IV infusion as per protocol specified dosing schedule.
  Other Names: MEDI2070
Drug: Brazikumab SC Injection — Brazikumab IV infusion as per protocol specified dosing schedule.
  Other Names: MEDI2070
Drug: Placebo — Placebo-matching Brazikumab IV infusion as per protocol specified dosing schedule.

SUMMARY:
A Phase 2b study to evaluate the efficacy and safety of brazikumab (MEDI2070) in participants with moderate to severe Crohn's disease who have failed or are intolerant to anti-tumor necrosis factor-alpha (anti-TNFα) therapy.

DETAILED DESCRIPTION:
This is a four-part Phase 2b study comprised of a 16-week, double-blind, placebo-controlled, Induction Period, a 12-week double-blind, placebo-controlled, Maintenance Period, a 24-week, Open-label Period and a post-treatment 28 week observational safety follow-up period designed to evaluate the short-term efficacy and the short- and long term safety of brazikumab in participants with moderate to severe, active Crohn's disease (CD) who have failed or are intolerant to anti-TNFα therapy as determined by the Investigator.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ileal, ileo-colonic, or colonic Crohn's Disease (CD) for > 3 months prior to screening
* Men or women age 18 - 80 years at the time of screening
* Moderate to severely active CD, as defined by Crohn's Disease Activity Index (CDAI) and endoscopic demonstration of inflammation
* Stable dose of medications for Crohn's disease therapy
* Prior treatment failure or intolerance with at least one Anti-Tumor Necrosis Factor-Alpha Therapy (anti-TNF α) agent
* Effective contraception from screening, and for 36 weeks after the last dose of investigational product
* No known history of active tuberculosis (TB) & negative assessment for TB/latent TB

Exclusion Criteria:

* Severe underlying immunosuppression
* Severe gastrointestinal complications; e.g., short bowel syndromes, obstructing strictures, recent or planned bowel surgery, Ileostomy and/or colostomy, recent bowel perforation
* Significant infections at screening; Infected abscess, positive for Clostridium difficile, recent infectious hospitalization
* Recent treatment with approved or investigational biologic therapy for Crohn's disease
* Recent or planned live attenuated vaccine
* History of cancer, except for basal cell carcinoma or carcinoma in situ (CIS) of the cervix with apparent cure ≥ 12 months before screening
* Pregnancy/breast feeding
* Drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-01-05 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2018-01-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (94):
- United States (51):
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Research Site, Phoenix, Arizona
  - South Denver Gastroenterology, PC, Lone Tree, Colorado
  - Research Site, Lone Tree, Colorado
  - Clinical Research of West Florida - Corporate, Clearwater, Florida
  - Borland-Groover Clinic, Jacksonville, Florida
  - Research Site, Jacksonville, Florida
  - Advanced Pharma CR, LLC, Miami, Florida
  - Research Site, Miami, Florida
  - IMIC, Inc., Palmetto Bay, Florida
  - Research Site, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Research Site, Evanston, Illinois
  - Indiana University, Indianapolis, Indiana
  - Research Site, Indianapolis, Indiana
  - Cotton-O'Neil Clinical Research Center, Digestive Health, Topeka, Kansas
  - Research Site, Topeka, Kansas
  - Graves Gilbert Clinic, Bowling Green, Kentucky
  - Research Site, Bowling Green, Kentucky
  - Research Site, Louisville, Kentucky
  - University of Louisville, Louisville, Kentucky
  - Clinical Trials of SW Louisiana, LLC, Lake Charles, Louisiana
  - Research Site, Lake Charles, Louisiana
  - Clinical Trials Management, LLC, Metairie, Louisiana
  - Research Site, Metairie, Louisiana
  - Research Site, Ann Arbor, Michigan
  - University of Michigan Health System, Ann Arbor, Michigan
  - Research Site, Southfield, Michigan
  - Revival Research Institute, LLC, Southfield, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Research Site, Rochester, Minnesota
  - Ehrhardt Clinical Research, LLC, Belton, Missouri
  - Research Site, Belton, Missouri
  - New York University Medical Center, Great Neck, New York
  - Premier Medical Group of the Hudson Valley, PC, Poughkeepsie, New York
  - Research Site, Poughkeepsie, New York
  - Research Site, Charlotte, North Carolina
  - Clinical Inquest Center Ltd, Dayton, Ohio
  - Research Site, Dayton, Ohio
  - Donald Guthrie Foundation, Sayre, Pennsylvania
  - Research Site, Sayre, Pennsylvania
  - Erlanger Health System, Chattanooga, Tennessee
  - Research Site, Chattanooga, Tennessee
  - Research Site, Houston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Gastroenterology Research of America, Houston, Texas
  - Baylor Research Institute, Temple, Texas
  - Research Site, Temple, Texas
  - Allegiance Research Specialists, LLC, Milwaukee, Wisconsin
  - Research Site, Wauwatosa, Wisconsin
- Australia (2):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Research Site, Woolloongabba
- Belgium (4):
  - Imeldaziekenhuis, Bonheiden
  - Research Site, Bonheiden
  - Research Site, Leuven
  - UZ Leuven, Leuven
- Canada (5):
  - London Health Science Centre, London, Ontario
  - Research Site, London, Ontario
  - LHSC - Victoria Hospital, London, Ontario
  - Research Site, Saskatoon, Saskatchewan
  - Royal University Hospital, Saskatoon, Saskatchewan
- France (8):
  - CHU de Toulouse - Hôpital Rangueil, Toulouse, Haute Garonne
  - CHU Rennes - Hôpital Pontchaillou, Rennes, Ille Et Vilaine
  - Hôpital de Brabois Adultes, Vandœuvre-lès-Nancy, Meurthe Et Moselle
  - CHU Saint Etienne - Hôpital Nord, Saint-Étienne-de-Montluc, Pays de la Loire Region
  - Research Site, Rennes
  - Research Site, Saint-Priez En Jarez
  - Research Site, Toulouse
  - Research Site, Vandœuvre-lès-Nancy
- Germany (4):
  - Medizinische Hochschule Hannover, Marburg, Hesse
  - St. Johannes Hospital, Dortmund, North Rhine-Westphalia
  - Research Site, Dortmund
  - Research Site, Hanover
- Hungary (4):
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Research Site, Budapest
  - Semmelweis Egyetem, Budapest
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
- Israel (2):
  - Kaplan Medical Center, Rehovot
  - Research Site, Rehovot
- Italy (2):
  - Istituto Clinico Humanitas, Rozzano, Milano
  - Research Site, Rozzano
- Netherlands (4):
  - Maastricht University Medical Center, Maastricht
  - Research Site, Maastricht
  - Erasmus Medisch Centrum, Rotterdam
  - Research Site, Rotterdam
- Russia (4):
  - Research Site, Krasnoyarsk
  - TSBIH "Territorial Clinical Hospital", Krasnoyarsk
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Research Site, Saint Petersburg
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Barcelona
  - Research Site, L'Hospitalet de Llobregat

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study enrolled 29 participants who were randomized to one of five treatment groups (Placebo/ Brazikumab High dose/ Brazikumab High-Medium dose/ Brazikumab Low dose/ Brazikumab Low-Medium dose). This study was terminated early.
Groups:
- Double Blind (DB): Placebo: Placebo-matching brazikumab intravenous (IV) infusion and subcutaneous (SC) injection at Weeks 0 and 4 followed by placebo-matching brazikumab SC injection at Weeks 8 and 12 in the induction phase and at Weeks 16, 20 and 24 in the maintenance phase.
- DB: Brazikumab High Dose: Brazikumab 700 mg, IV infusion and placebo-matching brazikumab, SC injection at Weeks 0 and 4 followed by brazikumab 210 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 210 mg, SC injection every 4 weeks at Weeks 8 and 12 in the induction phase and Weeks 16, 20 and 24 in the maintenance phase.
- DB: Brazikumab High-Medium Dose: Brazikumab 280 mg, IV infusion and placebo-matching brazikumab, SC injection at Week 0 followed by brazikumab 210 mg, SC injection and placebo-matching brazikumab IV infusion at Week 4, followed by brazikumab 210 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 210 mg, SC injection every 4 weeks up to Week 24 in the maintenance phase.
- DB: Brazikumab Low-Medium Dose: Brazikumab 210 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 0 followed by brazikumab 105 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 105 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 105 mg, SC injection every 4 weeks up to Week 24 in the maintenance phase.
- DB: Brazikumab Low Dose: Brazikumab 70 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 0 followed by brazikumab 35 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 35 mg, SC injection at Weeks 8 and 12 in the induction phase. Participants received brazikumab 35 mg, SC injection every 4 weeks up to Week 24 in the maintenance phase.
- Open-label (OL): Placebo/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received placebo-matching brazikumab in the double-blind treatment period.
- OL: Brazikumab High Dose/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received high dose of brazikumab in the double-blind treatment period.
- OL: Brazikumab High- Medium Dose/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received high-medium dose of brazikumab in the double-blind treatment period.
- OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received low-medium dose of brazikumab in the double-blind treatment period.
- OL: Brazikumab Low Dose/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received low dose of brazikumab in the double-blind treatment period.
Period: Double-blind Period
Arm/Group | Double Blind (DB): Placebo | DB: Brazikumab High Dose | DB: Brazikumab High-Medium Dose | DB: Brazikumab Low-Medium Dose | DB: Brazikumab Low Dose | Open-label (OL): Placebo/Brazikumab 210 mg | OL: Brazikumab High Dose/Brazikumab 210 mg | OL: Brazikumab High- Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low Dose/Brazikumab 210 mg
Started | 5 | 5 | 9 | 7 | 3 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 4 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 1 | 7 | 4 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Non-Compliance With Study Drug | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study Terminated By Sponsor | 1 | 1 | 5 | 2 | 2 | 0 | 0 | 0 | 0 | 0
Not completed — Reason Not Specified | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Open-label (OL) Period
Arm/Group | Double Blind (DB): Placebo | DB: Brazikumab High Dose | DB: Brazikumab High-Medium Dose | DB: Brazikumab Low-Medium Dose | DB: Brazikumab Low Dose | Open-label (OL): Placebo/Brazikumab 210 mg | OL: Brazikumab High Dose/Brazikumab 210 mg | OL: Brazikumab High- Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low Dose/Brazikumab 210 mg
Started | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 2 | 3 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Not completed — Study Terminated By Sponsor | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized into the study and received at least 1 whole dose of investigational product for the 28-week, double-blind, placebo-controlled treatment period.
Groups:
- Brazikumab High-Medium Dose: Brazikumab 280 mg, IV infusion and placebo-matching brazikumab, SC injection at Week 0 followed by brazikumab 210 mg, SC injection and placebo-matching brazikumab, IV infusion at Week 4, followed by brazikumab 210 mg, SC injection in the induction phase. Participants received brazikumab 210 mg, SC injection every 4 weeks in the maintenance phase and open-label period up to Week 48.
- Total: Total of all reporting groups
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose | Total
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.3 (10.34) | 37.2 (13.29) | 38.3 (15.03) | 39.9 (13.89) | 40.7 (11.37) | 38.3 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 6 | 4 | 1 | 16
  Male | 2 | 2 | 3 | 3 | 2 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 2
  Not Hispanic or Latino | 4 | 5 | 8 | 5 | 3 | 25
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1 | 0 | 2
  White | 3 | 5 | 8 | 6 | 3 | 25
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Remission at Week 8
Description: CDAI remission was defined as a CDAI score of <150 at Week 8. CDAI score was calculated by summing weighted scores for subjective items [number of liquid or very soft stools, abdominal pain (on a scale of 0=none to 3=severe) and general well-being (on a scale of 1=generally well to 4=terrible)] recorded by a diary during a 1-week period, and objective items [associated symptoms, taking antidiarrheal agents such as loperamide/opiates, abdominal mass, hematocrit, daily morning temperature, and body weight]. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Week 8
Population: ITT population included all participants who were randomized into the study and received at least 1 whole dose of investigational product for the 28-week, double-blind, placebo-controlled treatment period.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants | 0.0 | 0.0 | 22.2 | 0.0 | 33.3

2. Secondary Outcome: Percentage of Participants With Loose/Liquid Stool Frequency Response
Description: Loose/liquid stool frequency response is the stools identified as Type 6 or 7 on Bristol Stool Form Scale, ≥ 30% reduction in weekly loose/liquid stool count compared to baseline. The participant recorded their stool consistency each day in a daily patient diary using the Bristol Stool Form Scale. It is a scale between 1-7, it measured the shape of the stool, where 1 correlates with the firmest stool and 7 correlates with entirely liquid stool.
Time Frame: Baseline, Weeks 8, 16 and 28
Population: ITT population included all participants who were randomized into the study and received at least 1 whole dose of investigational product for the 28-week, double-blind, placebo-controlled treatment period. Participant with missing data for this outcome measure was imputed as a non-responder.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 50.0 | 40.0 | 55.6 | 14.3 | 66.7
  Week 16 | 50.0 | 60.0 | 66.7 | 0.0 | 33.3
  Week 28 | 25.0 | 20.0 | 33.3 | 0.0 | 33.3

3. Secondary Outcome: Percentage of Participants With Crohn's Disease Activity Index (CDAI) Response
Description: CDAI response was defined as a decrease from baseline in the CDAI score of ≥100. CDAI score was calculated by summing weighted scores for subjective items [number of liquid or very soft stools, abdominal pain (on a scale of 0=none to 3=severe) and general well-being (on a scale of 1=generally well to 4=terrible)] recorded by a diary during a 1-week period, and objective items [associated symptoms, taking antidiarrheal agents such as loperamide/opiates, abdominal mass, hematocrit, daily morning temperature, and body weight]. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Baseline, Weeks 8, 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 0.0 | 60.0 | 77.8 | 28.6 | 66.7
  Week 16 | 25.0 | 60.0 | 55.6 | 14.3 | 33.3
  Week 28 | 0.0 | 50.0 | 11.1 | 14.3 | 33.3

4. Secondary Outcome: Percentage of Participants With CDAI Clinical Remission
Description: CDAI clinical remission was defined as a CDAI score of <150. CDAI score was calculated by summing weighted scores for subjective items [number of liquid or very soft stools, abdominal pain (on a scale of 0=none to 3=severe) and general well-being (on a scale of 1=generally well to 4=terrible)] recorded by a diary during a 1-week period, and objective items [associated symptoms, taking antidiarrheal agents such as loperamide/opiates, abdominal mass, hematocrit, daily morning temperature, and body weight]. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 16 and 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 16 | 25.5 | 20.0 | 22.2 | 14.3 | 33.3
  Week 28 | 25.0 | 0.0 | 0.0 | 0.0 | 33.3

5. Secondary Outcome: Percentage of Participants With Simple Endoscopic Score for Crohn's Disease (SES-CD) Response
Description: SES-CD response was defined as a decrease from baseline in SES-CD score of ≥ 50%. The SES-CD evaluates 4 endoscopic variables [ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis] each rated from 0 (best) to 3 (worst) in 5 segments evaluated during ileocolonoscopy [ileum, right colon, transverse colon, left colon, and rectum]. The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 60, where higher scores indicates more severe disease.
Time Frame: Baseline, Weeks 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 16 | 0.0 | 40.0 | 44.4 | 14.3 | 0.0
  Week 28 | 0.0 | 40.0 | 11.1 | 14.3 | 33.3

6. Secondary Outcome: Percentage of Participants With Loose/Liquid Stool Frequency Remission
Description: as for outcome 2
Time Frame: Baseline, Weeks 8, 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 75.0 | 60.0 | 55.6 | 28.6 | 100.0
  Week 16 | 50.0 | 60.0 | 55.6 | 14.3 | 66.7
  Weeks 28 | 50.0 | 20.0 | 33.3 | 14.3 | 33.3

7. Secondary Outcome: Percentage of Participants With Simple Endoscopic Score for Crohn's Disease (SES-CD) Remission
Description: SES-CD remission was defined as a Total SES-CD score of ≤4 and no subscore >2. The SES-CD evaluates 4 endoscopic variables [ulcer size, proportion of the surface area that is ulcerated, proportion of the surface area affected, and stenosis] each rated from 0 (best) to 3 (worst) in 5 segments evaluated during ileocolonoscopy [ileum, right colon, transverse colon, left colon, and rectum]. The score for each endoscopic variable is the sum of values obtained for each segment. The SES-CD total is the sum of the 4 endoscopic variable scores from 0 to 60, where higher scores indicates more severe disease.
Time Frame: Weeks 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 16 | 0.0 | 20.0 | 22.2 | 0.0 | 0.0
  Week 28 | 0.0 | 20.0 | 11.1 | 0.0 | 0.0

8. Secondary Outcome: Percentage of Participants With Patient Response Outcome-2 (PRO2) Remission
Description: PRO2 evaluated 2 patient-reported symptoms: the frequency of liquid or soft stools and abdominal pain (on an 11-point scale where 0=no pain to 10=worst imaginable pain). A weekly score was calculated for the liquid or soft stool frequency and a separate weekly score was calculated for abdominal pain, in each case based on daily symptom reporting. PRO2-remission was defined as PRO2 less than 8 points. PRO2 is a composite index consisting of weighted scoring of both variables. PRO2 scores ranges from 0 to approximately 45, higher score indicates higher disease activity.
Time Frame: Weeks 8, 16 and 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 0.0 | 20.0 | 11.1 | 0.0 | 0.0
  Week 16 | 0.0 | 20.0 | 0.0 | 0.0 | 0.0
  Week 28 | 25.0 | 0.0 | 11.1 | 0.0 | 0.0

9. Secondary Outcome: Percentage of Participants With PRO2 Response
Description: PRO2 evaluated 2 patient-reported symptoms: the frequency of liquid or soft stools and abdominal pain. PRO2 response was defined as remission or response in one symptom (either abdominal pain or stool frequency) plus response in the other: a) abdominal pain remission: On an 11-point (0 to 10) pain scale: During 1 week, no daily score > 2, b) abdominal pain response: On an 11-point (0 to 10) pain scale: ≥ 30% reduction in weekly pain score from baseline, c) loose/liquid stool frequency remission: Counting stools identified as Type 6 or 7 on Bristol Stool Form Scale (BSFS), (The BSFS is a scale between 1-7, where 1 correlates with the firmest stool and 7 correlates with entirely liquid stool), during 1 week, each daily loose/liquid stool count ≤ 3, d) loose/liquid stool frequency response: Counting stools identified as Type 6 or 7 on BSFS, ≥ 30% reduction in weekly loose/liquid stool count compared to baseline.
Time Frame: Baseline, Weeks 8, 16 and 28
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 50.0 | 20.0 | 33.3 | 0.0 | 66.7
  Week 16 | 50.0 | 40.0 | 66.7 | 0.0 | 66.7
  Week 28 | 50.0 | 0.0 | 33.3 | 0.0 | 33.3

10. Secondary Outcome: Serum Interleukin (IL)-22 and Serum Lipocalin 2 (LCN2) Concentration as a Biomarker of Brazikumab's Efficacy
Time Frame: Weeks 16 and 28
Population: Data for predictive biomarker analysis was not collected due to small number of participants available for analysis.
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Percentage of Participants With CDAI Modified Sustained Clinical Remission at Both Weeks 8 and 28
Description: CDAI modified sustained clinical remission was defined as a CDAI score of <150 at both Weeks 8 and 28. CDAI score was calculated by summing weighted scores for subjective items [number of liquid or very soft stools, abdominal pain (on a scale of 0=mild to 3=severe) and general well-being (on a scale of 1=generally well to 4=terrible)] recorded by a diary during a 1-week period, and objective items [associated symptoms, taking antidiarrheal agents such as loperamide/opiates, abdominal mass, hematocrit, daily morning temperature and body weight]. CDAI scores range from 0 to approximately 600 points, higher score indicates higher disease activity.
Time Frame: Weeks 8 and 28
Population: Data was not collected for this endpoint.
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Serum Brazikumab Concentration
Time Frame: Predose at Weeks 0, 1, 4, 8, 12, 16, 28; Postdose at Weeks 0 and 4
Population: The Pharmacokinetic (PK) population included all participants who received at least 1 dose of investigational product and had at least 1 PK sample containing quantifiable brazikumab. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Mean (Standard Deviation); unit: nanograms per milliliters (ng/mL)
Arm/Group | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 5 | 9 | 7 | 3
nanograms per milliliters (ng/mL)
  Week 0, Predose | 307 (686) | 3213 (9639) | 7 (19) | 0 (0)
  Week 0, Postdose: number analyzed (Participants) | 4 | 7 | 6 | 3
  Week 0, Postdose | 448085 (151153) | 149388 (75443) | 0 (0) | 0 (0)
  Week 1, Predose | 124239 (19941) | 51335 (16422) | 20740 (10744) | 14073 (5896)
  Week 4, Predose: number analyzed (Participants) | 5 | 7 | 7 | 3
  Week 4, Predose | 56798 (25064) | 17741 (4622) | 11201 (6084) | 5290 (266)
  Week 4, Postdose: number analyzed (Participants) | 4 | 8 | 7 | 3
  Week 4, Postdose | 390820 (60355) | 17252 (10812) | 11383 (5853) | 7555 (4178)
  Week 8, Predose: number analyzed (Participants) | 5 | 9 | 6 | 3
  Week 8, Predose | 77747 (30129) | 13997 (4467) | 10850 (4191) | 7982 (5967)
  Week 12, Predose | 50667 (16704) | 19076 (11823) | 11554 (4505) | 6031 (3528)
  Week 16, Predose: number analyzed (Participants) | 5 | 7 | 5 | 3
  Week 16, Predose | 33247 (12890) | 26321 (16994) | 13920 (5340) | 6404 (1768)
  Week 28, Predose: number analyzed (Participants) | 2 | 2 | 3 | 1
  Week 28, Predose | 31067 (8738) | 13713 (2072) | 10842 (6641) | 6988 (NA) — Standard deviation (SD) was not estimable for one participant.

13. Secondary Outcome: Number of Participants With Serum Anti-drug Antibodies for Brazikumab
Time Frame: Predose at Weeks 0, 4, 12, 16, 28, 40 and 52
Population: ITT population included all participants who were randomized into the study and received at least 1 whole dose of investigational product for the 28-week, double-blind, placebo-controlled treatment period. Number analyzed is number of participants with evaluable data at given time-point.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
Participants
  Week 0 | 0 | 1 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 4 | 5 | 8 | 7 | 3
  Week 4 | 0 | 0 | 1 | 0 | 0
  Week 12 | 0 | 1 | 0 | 0 | 0
  Week 16: number analyzed (Participants) | 3 | 5 | 6 | 4 | 3
  Week 16 | 0 | 0 | 0 | 0 | 0
  Week 28: number analyzed (Participants) | 2 | 2 | 3 | 3 | 1
  Week 28 | 0 | 0 | 0 | 0 | 0
  Week 40: number analyzed (Participants) | 2 | 1 | 3 | 2 | 0
  Week 40 | 0 | 0 | 0 | 0 |
  Week 52: number analyzed (Participants) | 0 | 1 | 3 | 1 | 0
  Week 52 |  | 0 | 0 | 0 |

14. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Treatment Emergent Serious Adverse Events (TESAEs), TEAEs of Special Interest and TEAEs Leading to Discontinuation
Description: An AE is any untoward medical occurrence in a patient/clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with treatment. An adverse event can therefore be any unfavorable and unintended sign (including abnormal laboratory finding), symptom, or disease temporally associated with the use of investigational product, whether or not related to the investigational product. A TEAE is any new AE or worsening of an existing condition after initiation of treatment. An SAE is an AE that resulted in death, inpatient hospitalization/prolongation of existing hospitalization, persistent or significant disability or incapacity, life threatening, a congenital anomaly/birth defect, or an important medical event. AE of special interest were infusion/injection-site reactions, hypersensitivity reactions, malignancies, cardiac events like myocardial infarction, stroke/cardiovascular death, ocular AE including cataracts.
Time Frame: From first dose of study drug up to 28 weeks post last dose (approximately up to Week 80)
Population: Safety population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 5 | 5 | 9 | 7 | 3
Participants
  TEAEs | 5 | 4 | 8 | 7 | 2
  TESAEs | 0 | 1 | 0 | 2 | 1
  TEAEs of Special Interest | 0 | 0 | 0 | 1 | 1
  TEAEs Leading to Discontinuation | 1 | 0 | 0 | 1 | 0

15. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Values
Description: Laboratory parameters included tests for hematology, serum chemistry and urinalysis. Laboratory values that were outside the reference range, considered clinically significant were reported.
Time Frame: From first dose of study drug up to 28 weeks post last dose (approximately up to Week 80)
Population: Safety population included all participants who received at least 1 dose of investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 5 | 5 | 9 | 7 | 3
Participants | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Percentage of Participants With Abdominal Pain Response
Description: Abdominal pain response is defined as a ≥ 30% reduction in weekly pain score from baseline on an 11-point (0 to 10) pain scale, where 0 = no pain and 10 = worst imaginable pain.
Time Frame: Baseline; Weeks 8, 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 50.0 | 40.0 | 44.4 | 28.6 | 66.7
  Week 16 | 50.0 | 60.0 | 66.7 | 28.6 | 100.0
  Week 28 | 50.0 | 0.0 | 33.3 | 0.0 | 33.3

17. Secondary Outcome: Percentage of Participants With Abdominal Pain Remission
Description: Abdominal pain remission is defined as no daily score > 2 on an 11-point (0 to 10) pain scale during 1 week, where 0 = no pain and 10 = worst imaginable pain.
Time Frame: Weeks 8, 16 and 28
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Brazikumab High Dose | Brazikumab High-Medium Dose | Brazikumab Low-Medium Dose | Brazikumab Low Dose
Number analyzed (Participants) | 4 | 5 | 9 | 7 | 3
percentage of participants
  Week 8 | 0.0 | 20.0 | 11.1 | 0.0 | 0.0
  Week 16 | 0.0 | 40.0 | 0.0 | 0.0 | 0.0
  Week 28 | 25.0 | 0.0 | 11.1 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 28 weeks post last dose (approximately up to Week 80)
Description: Safety population included all participants who received at least 1 dose of investigational product.
Groups:
- DB: Placebo: Placebo-matching brazikumab intravenous (IV) infusion and subcutaneous (SC) injection at Weeks 0 and 4 followed by placebo-matching brazikumab SC injection at Weeks 8 and 12 in the induction phase and at Weeks 16, 20 and 24 in the maintenance phase.
- OL: Placebo/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received placebo-matching brazikumab in the double-blind treatment period.
- OL: Brazikumab High-Medium Dose/Brazikumab 210 mg: Brazikumab 210 mg, SC injection every 4 weeks in the open-label period starting at Week 28 up to Week 48. Participants received high-medium dose of brazikumab in the double-blind treatment period.
Arm/Group | DB: Placebo | DB: Brazikumab High Dose | DB: Brazikumab High-Medium Dose | DB: Brazikumab Low-Medium Dose | DB: Brazikumab Low Dose | OL: Placebo/Brazikumab 210 mg | OL: Brazikumab High Dose/Brazikumab 210 mg | OL: Brazikumab High-Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg | OL: Brazikumab Low Dose/Brazikumab 210 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/9 | 0/7 | 0/3 | 0/2 | 0/3 | 0/2 | 0/3 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/5 | 0/9 | 1/7 | 1/3 | 0/2 | 0/3 | 0/2 | 1/3 | 0/1
Other Adverse Events (participants affected / at risk) | 5/5 | 4/5 | 8/9 | 7/7 | 1/3 | 2/2 | 1/3 | 1/2 | 1/3 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=5) | DB: Brazikumab High Dose (N=5) | DB: Brazikumab High-Medium Dose (N=9) | DB: Brazikumab Low-Medium Dose (N=7) | DB: Brazikumab Low Dose (N=3) | OL: Placebo/Brazikumab 210 mg (N=2) | OL: Brazikumab High Dose/Brazikumab 210 mg (N=3) | OL: Brazikumab High-Medium Dose/Brazikumab 210 mg (N=2) | OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg (N=3) | OL: Brazikumab Low Dose/Brazikumab 210 mg (N=1)
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB: Placebo (N=5) | DB: Brazikumab High Dose (N=5) | DB: Brazikumab High-Medium Dose (N=9) | DB: Brazikumab Low-Medium Dose (N=7) | DB: Brazikumab Low Dose (N=3) | OL: Placebo/Brazikumab 210 mg (N=2) | OL: Brazikumab High Dose/Brazikumab 210 mg (N=3) | OL: Brazikumab High-Medium Dose/Brazikumab 210 mg (N=2) | OL: Brazikumab Low-Medium Dose/Brazikumab 210 mg (N=3) | OL: Brazikumab Low Dose/Brazikumab 210 mg (N=1)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Iritis (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal mycotic infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Postoperative abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eye naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0
Phlebitis superficial (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Drug intolerance (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Enterobiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Iron deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to small number of participants,29 randomized by study termination, only descriptive statistics for limited efficacy endpoints were provided. Enrollment did not achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/37/NCT02574637/Prot_SAP_000.pdf